CLINICAL TRIAL: NCT07194369
Title: Validation of the Setswana Translated Quality of Recovery Questionnaire in Orthopaedic Patients at a Tertiary Hospital in South Africa: a Cross-Sectional Observational Study
Brief Title: Validation of the Setswana Translated Quality of Recovery Questionnaire in Orthopaedic Patients at a Tertiary Hospital in South Africa
Status: Not yet recruiting | Type: Observational
Sponsor: Sefako Makgatho Health Sciences University (Other)
Responsible Party: Principal Investigator, Unathi Mzinyathi, DR, Sefako Makgatho Health Sciences University
Other Study IDs: SMUREC/M/276/2025:PG
Record Dates: First submitted 2025-09-01; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Quality of Recovery (QoR-15); Quality of Recovery From Anaesthesia
Keywords: Setswana translated QoR-15; Quality of Recovery in patients undergoing orthopaedic surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to evaluate the validity, reliability and feasibility of the Setswana-translated version of the 15-item Quality of Recovery (QoR-15) questionnaire. The question it aims to answer is:

Does the Setswana translation of the QoR-15 serve as a valid, reliable and user friendly tool for assessing postoperative recovery in Setswana speaking patients undergoing orthopaedic surgery at a tertiary hospital in Gauteng, South Africa?

The participants will be asked to complete the Setswana-translated QoR-15 questionnaire both preoperatively and postoperatively.

In addition, they will be asked to rate their overall postoperative recovery using a visual analog scale (VAS).

DETAILED DESCRIPTION:
Patient reported outcome measures are increasingly recognised as important in preoperative research, yet their routine use in clinical practice remains limited in South Africa.

While quality of recovery measures have been widely applied in general and ambulatory surgery settings, there is a relative paucity of data specifically addressing orthopaedic populations.

Orthopaedic surgical procedures are associated with significant postoperative pain, functional limitations and extended rehabilitation periods, all of which can substantially impact the patient's overall recovery experience. Evaluating a short-term postoperative outcome like quality of recovery in this surgical cohort may help tailor postoperative care to patient needs, which may lead to better patient-clinician communication, better surgical outcomes and better patient satisfaction.

A lack of standardised and validated outcome measures in local languages and high rates of illiteracy may be impediments to implementing widespread use of patient reported outcome questionnaires in practice. Patients who are functionally literate may still not understand medical terms if not presented in their home language and proficiency in English varies widely across South Africa. South Africa has a diverse language heritage with 11 official languages and high rates of functional illiteracy. While many South Africans are able to communicate in English, only a small minority reports English as the primary language used most often outside the household. For black South Africans, the most common languages spoken outside of the home most commonly are IsiZulu, IsiXhosa and the Sotho-Tswana languages.

At present, validated translations of the QoR-15 questionnaire are only available in English and IsiZulu for South African use.

By adding another validated translation in a local language, it is hoped that it will be easier to measure quality of recovery in Setswana speaking populations to address health disparities.

A Setswana translation of the QoR-15 questionnaire exists from a previous study which may be of use in Ga-Rankuwa, which is home to a Setswana speaking population. This translated questionnaire is yet to be validated in this population. For patient reported outcome measures (PROMs) to be effective in non-English speaking populations, rigorous linguistic and cultural adaptation is necessary.

In this study, quality of recovery will be measured with the Setswana translation of the QoR-15 questionnaire as well as with a visual analog scale on which patients can rate their overall postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* Scheduled elective orthopaedic surgery at Dr George Mukhari Academic Hospital

Exclusion Criteria:

* Patients who are not fluent in Setswana
* Patients booked for emergency surgery where a delay to surgery could be detrimental.
* Patients where the surgery is delayed beyond 10 days of the initial assessment and pre-operative QoR-15 measurement.
* Patients with a psychiatric disturbance that precludes complete co-operation.
* Patients with a severe debilitating medical or surgical condition that may limit objective assessment after surgery.
* Patients with any life threatening postoperative complication.
* Postoperative confusion or delirium.
* Patients with a history of recent drug or alcohol abuse which may render responses unreliable.
* Incomplete QoR-15 questionnaires.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (aged 18 years and older) who are fluent in Setswana and are scheduled for elective orthopaedic surgery at the hospital. The population is expected to be diverse in terms of gender, age, and socioeconomic background, reflecting the typical demographic of Setswana-speaking patients. These patients are expected to be conscious and alert in the postoperative period, able to provide informed consent, and cognitively capable of understanding and responding to a questionnaire. Participants with known cognitive impairments, severe postoperative complications that impair communication, or those unwilling to participate will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Convergent validity of the Setswana-translated QoR-15 score | Pre-operative baseline and 24 hours postoperatively.
  To evaluate convergent validity by assessing the Spearman correlation between the Setswana-translated QoR-15 score and a general visual analog scale (VAS).
  Unit of measure: Correlation co-efficient (r).

SECONDARY OUTCOMES:
Construct validity of the Setswana-translated QoR-15 score | Pre-operative (baseline) and 24 hours postoperatively
  To evaluate construct validity by assessing associations between the QoR-15 score and patient factors (age, gender, duration & severity of surgery).
  Unit of Measure: Regression coefficients/association statistics
Internal consistency of the Setswana translated QoR-15 score | Pre-operative (baseline) and 24 hours postoperatively
  To evaluate internal consistency using Cronbach's alpha based on the average correlation between the QoR-15 items.
Test-retest variability of the Setswana-translated QoR-15 score | 60 minutes after first postoperative questionnaire
  To evaluate test-retest variability in a subset of 25 patients who will be asked to complete a repeat assessment 60 minutes after their first postoperative questionnaire.
  Unit of measure: intraclass correlation coefficient
Acceptability and feasibility of the Setswana-translated QoR-15 score | During recruitment and postoperative assessment
  To evaluate acceptability and feasibility by calculating the recruitment rate, completion rate and time taken to complete the questionnaire
Responsiveness of the Setswana-translated QoR-15 score | Pre-operative (baseline) and 24 hours postoperatively.
  To evaluate responsiveness by calculating Cohen's effect size of change in QoR-15 scores from pre-operative to postoperative assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Charle Dr Steyl, Study Director — Sefako Makgatho Health Sciences University
Locations (1):
- Dr George Mukhari Academic Hospital, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No
Regarding anonymity of patient information, the only documents to contain the patient's name will be the consent form and a sequentially numbered list that will be completed at recruitment that the PI will store to keep track of patients in the study. All data will be de-identified, no personal information (for example name and file number) will be recorded on any of the other study documents.
  Confidentiality will be ensured by the PI storing all paper documents in lever-arch files in a secure location that only the PI and research assistant has access to. The sequentially numbered list will be stored electronically in a password controlled online folder that only the PI has access to. Personal information will not be shared without express patient permission.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT07194369/Prot_SAP_ICF_000.pdf